CLINICAL TRIAL: NCT03455569
Title: A Dyadic Sleep Intervention for Alzheimer's Disease Patients and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Yeonsu Song, PhD, RN, FNP, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1K23AG055668-05 (NIH)
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Sleep; Alzheimer Disease
Keywords: Behavioral sleep management; Alzheimer's disease; Informal caregiver
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral sleep education (Experimental): manual-based sleep hygiene recommendations and a behavioral sleep intervention including sleep compression therapy
  Interventions: Behavioral: Behavioral sleep education
- Education only (Experimental): education on sleep, aging, and dementia but without specific or individualized recommendations
  Interventions: Behavioral: Education only

INTERVENTIONS:
Behavioral: Behavioral sleep education — This group will receive manual-based sleep hygiene recommendations and a behavioral sleep intervention including sleep compression therapy
  Arms: Behavioral sleep education
Behavioral: Education only — This group will receive information about sleep, aging, and dementia, but without specific or individualized recommendations
  Arms: Education only

SUMMARY:
Studies consistently show the negative health impact of sleep problems in both Alzheimer's disease (AD) patients and their caregivers. However, only a few sleep interventions have been conducted for AD patients or their caregivers in community settings and none have addressed both members of the dyad concurrently. To fill these gaps, this study aims to develop a sleep intervention program specifically tailored for AD patient/caregiver dyads who both experience sleep difficulties.

DETAILED DESCRIPTION:
In 2015, Americans provided 18 billion hours of unpaid care for patients with Alzheimer's disease (AD) and other dementias, with an economic value of $221 billion. This estimate may be even higher among caregivers of AD patients when they have sleep problems. In fact, the caregivers' sleep is often disturbed by nighttime sleep disturbance of AD patients, which is one of the major reasons why those patients are admitted to institutions. Due to the bidirectional nature of sleep disturbance in AD patients and their caregivers, it is critical to develop a sleep intervention program for the dyad that addresses sleep disturbance in both individuals.

Nighttime sleep disturbance in AD patients is associated with shorter survival, lower quality of life, and decreased social engagement. Poor sleep among their caregivers is associated with increased depressive symptoms, higher levels of caregiver role burden, and increased inflammation, which is known to increase risk for cardiovascular disease. Such decline in caregivers' health may then impact the quality of care for AD patients.

Behavioral sleep intervention programs for AD patients or caregivers are feasible but long-term effects on improving sleep and health remain unclear. No behavioral sleep interventions have focused on the patient-caregiver dyad, and only a few behavioral sleep intervention studies have targeted community-dwelling AD patients or caregivers. Dyad-based sleep interventions may have better effects on sleep and other health outcomes because of the influence of AD patients on their caregivers and vice versa.

The proposed intervention focuses on educating caregivers to improve their own and the patients' sleep, using behavioral sleep management techniques. This intervention builds upon a previous caregiver focus group study (VA HSR&D LIP 65-154, PI: Song) and the existing sleep interventional research studies, which included patients with mild cognitive impairments and AD patients. The sleep program involves 4 face-to-face meetings plus 1 telephone session. Phase 1 study aims to iteratively refine and finalize the intervention program materials with 5 AD patient/caregiver dyads. Phase 2 study aims to pilot test the effects of the intervention program (n=20 dyads) on sleep, health, and quality of life in both members of the group, compared to a non-directive education-only control program (n=20 dyads) in a small randomized controlled trial. Primary outcomes will include objective sleep efficiency and total wake time measured by actigraphy for AD patients and subjective sleep measured by the Pittsburgh Sleep Quality Index for caregivers. A unique aspect of the proposed study is that the program is tailored to address sleep problems of both patients and caregivers, and includes upstream biomarkers to evaluate a key mechanism of intervention benefits that can be further explored in future research.

ELIGIBILITY:
Inclusion Criteria for Alzheimer's disease (AD) patients:

* AD diagnosis OR probable or possible AD as documented in electronic medical record, which includes Mini Mental State Exam score >12 (indicating mild to moderate severity of AD) and neuroimaging evidence
* Community-dwelling
* >1 sleep problem >3x/week on the Neuropsychiatric Inventory Nighttime Behavior Scale
* Aged >60 years
* Able to ambulate with or without assistive device
* Have an eligible caregiver (see below)

Inclusion Criteria for caregivers:

* Live with an eligible patient
* Aged >21 years
* Have regularly assisted patient with >1 of 6 basic activities of daily living (ADLs) (i.e., bathing, dressing, toileting, transfers, continence, feeding) or >1 of 8 Instrumental ADL (IADLs) (i.e., using the telephone, shopping, preparing meals, housekeeping, laundry, transportation, taking medicine, managing money) for the past 6 months
* Pittsburgh Sleep Quality Index (PSQI) total score >5
* Montreal Cognitive Assessment (MoCA) score >= 23
* Can communicate in English

Exclusion Criteria:

- If AD patient is bed bound

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency for Alzheimer's disease patients | 3 months after the last session of the sleep intervention
  Sleep efficiency (mean percent time asleep while in bed) will be calculated from 3 days of wrist actigraphy
Total wake time for Alzheimer's disease patients | 3 months after the last session of the sleep intervention
  Total wake time (mean total minutes awake from sleep onset to get up time) will be calculated from 3 days of wrist actigraphy
Sleep quality for caregivers | 3 months after the last session of the sleep intervention
  Total score on the Pittsburgh Sleep Quality Index will be used as a measure of sleep quality

SECONDARY OUTCOMES:
Cognitive function for Alzheimer's disease patients | 3 months after the last session of the sleep intervention
  Total score on the Alzheimer's Disease Assessment Scale-Cognitive Subscale test will be used as a measure of cognitive function
Problematic behaviors for Alzheimer's disease patients | 3 months after the last session of the sleep intervention
  Total score on the Revised Memory and Behavior Problem Checklist will be used as a measure of problematic behaviors
Depression for Alzheimer's disease patients | 3 months after the last session of the sleep intervention
  Total score on the Cornell Scale for Depression in Dementia will be used as a measure of depression
Caregiver burden for caregivers | 3 months after the last session of the sleep intervention
  Total score on the Zarit Burden Interview will be used as a measure of caregiver burden
Stress for caregivers | 3 months after the last session of the sleep intervention
  Total score on the Perceived Stress Scale will be used as a measure of stress
Depression for caregivers | 3 months after the last session of the sleep intervention
  Total score on the Center for Epidemiological Study-Depression will be used as a measure of depression
Inflammation for caregivers | 3 months after the last session of the sleep intervention
  Levels of C-reactive protein and gene expression of inflammation will be measured
Quality of life for Alzheimer's disease patients | 3 months after the last session of the sleep intervention
  Total score on the Quality of Life-Alzheimer's Disease Scale will be used as a measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yeonsu Song, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Veterans Affairs Greater Los Angeles Healthcare System, North Hills, California

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the primary outcome is published

REFERENCES:
- [Derived] Song Y, Papazyan A, Lee D, Mitchell MN, McCurry SM, Irwin MR, Teng E, Alessi CA, Martin JL. The feasibility of a sleep education program for informal dementia care dyads: A pilot randomized controlled trial. J Am Geriatr Soc. 2024 Apr;72(4):1207-1215. doi: 10.1111/jgs.18720. Epub 2024 Jan 9. PMID 38193336